CLINICAL TRIAL: NCT05941572
Title: Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) in Patients With Major Trauma and Uncontrolled Haemorrhagic Shock: a Retrospective Analysis
Brief Title: Resuscitative Endovascular Balloon Occlusion of the Aorta in Haemorrhagic Shock
Status: Withdrawn | Type: Observational
Why Stopped: change of study plan
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 35-345 ex 22/23
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2023-09

CONDITIONS: Non-compressible Torso Hemorrhage; Trauma Injury
Keywords: uncontrollable hemorrhage; trauma; ballon occlusion of the aorta
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Resuscitative endovascular balloon occlusion of the aorta (REBOA) is a procedure that has the goal to stabilize trauma patients with non-compressible torso hemorrhage by temporarily occluding the aorta with a ballon catheter to increase central perfusion and stop uncontrollable bleeding from the diaphragm downwards.

The investigators are planning to evaluate all patients who had a REBOA catheter placed at their clinic or in the pre-clinical setting from the start of 2019 to the 31.12.2022 who were transferred to their clinic, with basic demographic and clinical data, the procedural specifics, and their potential complications.

DETAILED DESCRIPTION:
Resuscitative endovascular balloon occlusion of the aorta (REBOA) is a procedure that has the goal stabilize trauma patients with non-compressible torso hemorrhage by temporarily occluding the aorta with a ballon catheter to increase central perfusion and stop uncontrollable bleeding from the diaphragm downwards.

The investigators plan to evaluate all patients who had a REBOA catheter placed at their clinic or in the pre-clinical setting from the start of 2019 to the 31.12.2022 who were transferred to their clinic, with basic demographic and clinical data, the procedural specifics, and their potential complications.

Investigators will search for patients who had a REBOA catheter placed in the study period in the clinical documentation system (openMEDOCS) and the database of the German trauma registry. Documentation will include hemodynamic parameters, transfused blood products, complications, basic demographics and mortality up to thirty days after REBOA placement.

The investigators will then try to find patients with similar trauma mechanism and severity of trauma in the German trauma registry and match them with their REBOA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-compressible torso hemorrhage following major trauma with REBOA placement
* age>18 years
* REBOA placement during the initial resuscitation

Exclusion Criteria:

* age<18 years
* missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients with non-compressible torso hemorrhage and REBOA placement in the initial resuscitation phase.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  all cause mortality
Occurrence of complications | 30 days
  Complications due to ballon occlusion of the aorta
Blood products | initial resuscitation phase (day one after admission)
  Used blood products

SECONDARY OUTCOMES:
hemodynamic improvement (blood pressure) | initial resuscitation phase (day one after admission)
  hemodynamic improvement after ballon occlusion of the aorta (blood pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Honnef, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria